CLINICAL TRIAL: NCT05214144
Title: The In4M Study: Integrating 4 Methods to Assess Physical Function in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2000031319; 2U01FD005938-03 (FDA)
Record Dates: First submitted 2022-01-13; First posted 2022-01-28 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Physical Function; Cancer, Breast; Lymphoma; Patient Empowerment; Patient Education; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Lymphoma; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- evaluating sources of physical function (PF): evaluate 4 distinct modalities of sources of PF (PRO, ClinRo, PerfO and wearable device data) on Hugo Health platform in breast cancer and lymphoma patients undergoing cytotoxic chemotherapy.
  Interventions: Other: PRO Instruments assessment questionnaire; Other: Baseline Survey Clinician- reported (ClinRO) ECOG; Device: Fitbit; Other: Hugo Health ("Hugo"); Other: 6 Minute Walk Test (6MWT)

INTERVENTIONS:
Other: PRO Instruments assessment questionnaire — Patient Reported Outcome (PRO) questionnaire consisting of:
  * PRO-CTCAE (approximately 11 questions plus free text)
  * Patient-Reported Outcomes Measurement Information System (PROMIS) physical function short form (version 8c) (8 questions)
  * PRO ECOG question (1 question)
  * EORTC Quality of Life questionnaire (QLQ)-F17 questions (17 questions)
  * Functional Assessment of Cancer Therapy-General version, rated on a 5-point Likert scale, (FACT-GP5) (single item global side effect bother question) (1 question)
  * The Patient Global Impression (PGI)-C and PGI-S items (anchors for physical function) (2 questions)
Other: Baseline Survey Clinician- reported (ClinRO) ECOG — Baseline Survey completed prior to initiation of chemotherapy
Device: Fitbit — wearable device
Other: Hugo Health ("Hugo") — an electronic platform that aggregates real world EHR data with patient's wearable and PRO data
Other: 6 Minute Walk Test (6MWT) — A comprehensive performance measure of exercise capacity, encompassing components of mobility, endurance, and functional capacity measure (PerfO)

SUMMARY:
This is a prospective observational cohort study. Breast cancer and lymphoma patients planned to receive cytotoxic therapy will be recruited at Yale and Mayo Clinic. The Study Period is 9 months, during which enrolled patients will use their personal smartphone, computer, or other web-connected device to connect with the Hugo platform which will deliver PRO questionnaires, and sync to the wearable device in the study (Fitbit). The PerfO (6MWT) will be conducted twice in clinic during the study period. Structured information from the electronic health record (EHR) and patient portals will be collected and where needed, the EHR will be directly reviewed to record AEs, hospitalizations/emergency department visits and dose delay/reductions. Required in-person face to face visit is only at baseline for consent, enrollment and receipt of wearable device; patients can be followed remotely afterward (i.e. do not need to be treated at Mayo or Yale)

DETAILED DESCRIPTION:
The purpose of this prospective observational study is to collect and evaluate 4 different sources of physical functioning (PF) data over the course of systemic anti-cancer therapy in lymphoma and breast cancer patients: clinician-reported Performance Status (PS), Patient Reported Outcomes (PROs), a Performance Outcome (PerfO) and patient wearable device data.

Aim 1: To measure PF using 4 distinct modalities (ClinRo, PRO, PerfO and wearable device data) on Hugo platform

* Characterize assessment challenges by comparing levels of missing data and reasons for missingness across the PF modalities
* Report on trajectories of function as ascertained by the 4 PF modalities

Aim 2: To explore associations between various sources of physical function data and determine change thresholds

* To identify measurement characteristics of the PF modalities including sensitivity to change and identification of meaningful change thresholds
* Compare change over time in data within and between the PF modalities
* Explore associations between changes in the various PF modalities and subsequent patient-reported adverse events (AEs), acute care use (unplanned hospitalizations or emergency department visits), other patient-reported domains of Health Related Quality of Life (HRQOL), and dose delay/reduction

Aim 3: To assess patient acceptability and experience using the different PF assessment modalities

• Administer an exit questionnaire to understand burden and usability of electronic PROs and wearable device data collection from the patient perspective

The allocation for patient recruitment is 18 months, with 9 months for follow up for each patient. The proposed overall project timeline is 3.5 years/39 months. A total of 200 patients will be enrolled at Yale Cancer Center and the Mayo Clinic, as outlined below. Data will be cleaned, reviewed, and analyzed as it is received from the Hugo platform on a rolling basis. Data analysis will be conducted at Mayo Clinic and Yale. Only de-identified data will be provided to the FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and over;
2. English- or Spanish-speaking;
3. Pregnant and non-pregnant patients are eligible for participation in this study
4. Eligible cancer type and planned intravenous cytotoxic chemotherapy regimen (defined as including 1 or more cytotoxic agents)
5. ECOG Performance Score of < 3
6. Breast cancer patients

   a) Patients with any stage breast cancer for whom a new intravenous cytotoxic chemotherapy regimen is planned within the next 8 weeks (patients with local/regional/distant recurrences are allowed; patients with concurrent/prior/future immunotherapy/radiotherapy, targeted therapy, and endocrine therapy for breast cancer are allowed)
7. Lymphoma patients

   a) Lymphoma patients of any histology, stage or line of treatment planned to receive a new intravenous cytotoxic containing chemotherapy regimen (patients planned to receive radiation, maintenance chemotherapy, consolidation stem cell transplant or chimeric antigen receptor T (CAR-T) cell therapy are allowed)
8. If patients are receiving the above standard therapies as part of a clinical trial which may include a novel agent or combination, they are also eligible for the present study if the therapeutic protocol permits enrollment in both studies
9. Willing and able to give consent and participate in study
10. Able to access a mobile device (smartphone or tablet) or computer with web access every day to complete study surveys; able to regularly upload data from the Fitbit to a device in a way that it can be transferred to Hugo
11. Willing and able to perform an in-clinic 6-minute walk test (gait aides are permitted if regularly used by the patient). If a patient is recruited remotely outside of Mayo Clinic Rochester or Yale Smilow Cancer Center New Haven, 6-minute walk test may be omitted.
12. Willing to use the health data sharing platform Potential subjects who do not meet all of the enrollment criteria will not be enrolled. Any deviations from these criteria must be reported in accordance with IRB Policies and Procedures.

Exclusion Criteria

1. Prior intravenous cytotoxic chemotherapy within 3 weeks prior to study enrollment
2. Excluded regimens (due to length of hospitalization required for chemotherapy administration):

   1. R-CODOX-M/IVAC,
   2. DA-R-EPOCH (inpatient)
3. Excluded histology (due to length of hospitalization and inpatient predominant treatment for required chemotherapy): primary central nervous system lymphoma

   a) Other regimens with an anticipated high duration of inpatient care time, at PI discretion
4. Lack of access to a mobile device (smartphone or tablet) or computer with web access
5. Unable or unwilling to connect Fitbit to device
6. Unable or unwilling to use the health data sharing platform
7. Unable to give consent and be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred patients will be recruited from two main sites: Yale and Mayo Clinic Rochester. Patient sampling will be stratified by site enrolled and cancer type. The investigator will seek to optimize diversity of the patient sample. Race/ethnicity will be determined by participant self-report, offering the opportunity for participants to select multiple races. Participants who self-define as part of a racial or ethnic minority and as white will be classified by their non-white race/ethnicity for purposes of counting enrollment quotas. The project team (including representatives from the FDA) will evaluate the enrollment throughout the study both in terms of counts as well as demographic mix. For the purposes of this study, specific goals or quotas are not being set.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
To measure Physical Function using Clinician Reported Outcomes (ClinRo) at baseline. | baseline
  ClinRo score at baseline using the Eastern Cooperative Oncology Group (ECOG) performance scale. Possible scores range from 0 to 5. The lower the score the better the performance.
Change in Patient Reported Outcomes Questionnaire: PRO-CTCAE | baseline, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, and Month 9.
  PRO-CTCAE is a patient-reported outcome (PRO) measurement system of 11 questions plus free text developed to evaluate symptomatic toxicity in patients on cancer clinical trials. Outcome reported as a count of adverse events.
Change in Patient Reported Outcomes Questionnaire: PROMIS | baseline, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, and Month 9.
  Patient-Reported Outcomes Measurement Information System (PROMIS), version 8c, is a patient reported survey which evaluates a patient physical function before and during treatment. It consists of 8 questions each scored from 5 (without any difficulty) to 1 (Unable to do).
Change in Patient Reported Outcomes Questionnaire: PRO ECOG | baseline, Week 2, Week 4, Week 6, Week 8, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, and Month 9.
  PRO ECOG is 1 question where patients describe their activity in the past month. Score ranges from 0 (normal with no limitations) to 3 (unable to perform activities, very limited).
Change in Patient Reported Outcomes Questionnaire: EORTC Quality of Life (QLQ)-F17 | baseline, Week 2, Week 4, Week 6, Week 8, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, and Month 9.
  EORTC Quality of Life questionnaire (QLQ)-F17 is a 17 question survey. The first 15 questions assess the patient's physical function and are scored from 1 (Not at all) to 4 (Very much). The final 2 questions asses the patient overall health and overall quality of life. Scoring ranges from 1 (very poor health/quality of life) to 7 (excellent health/quality of life).
Change in Patient Reported Outcomes Questionnaire: FACT-GP5 | baseline, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, and Month 9.
  Functional Assessment of Cancer Therapy-General version (FACT-GP5) is a single question in which patients report their bother by side effects of treatment. Scores range from 0 (not at all bothered by side effect) to 4 (very much bothered by side effects).
Change in Patient Reported Outcomes Questionnaire: Patient Global Impression-Change (PGI-C) and Patient Global Impression-Severity (PGI-S) | baseline, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, and Month 9.
  A two question survey. Question one, PGI-S, describes severity of symptoms of on a scale from 1 (normal severity) to 4 (severe symptoms). Question two, PGI-C, patients report how their physical function has changed from baseline on a scale from 1 (very much improved) to 7 (very much worse).
Change in Physical Function using Performance Outcome 6-Minute Walk Test | baseline and 3 months
  Performance Outcome measured using a 6-minute walk test. The outcome is distance in meters traveled by the patient in a 6 minute time period at baseline and 3 months to evaluate patient performance before and after chemotherapy.
Steps Data From Wearable Device | baseline through month 9
  Count of total daily steps and maximum cadence (steps/minute) with activity data collected using a Fitbit at baseline (7 days prior to the start of chemotherapy) continually until Month 9.
Heart Rate Data From Wearable Device | baseline through month 9
  Resting heart rate (beats/minute) and heart rate during moderate to vigorous physical activity (MVPA) data collected using a Fitbit at baseline (7 days prior to the start of chemotherapy) continually until Month 9.
Patient Activity Data From Wearable Device | baseline through month 9
  Daily duration of MVPA (in minutes), count of ≥10-minute bouts of MVPA, daily duration of sedentary time (in minutes), and count of ≥ 10-minutes bouts of sedentary time (in minutes) data collected using a Fitbit at baseline (7 days prior to the start of chemotherapy) continually until Month 9.

CONTACTS AND LOCATIONS:
Overall Officials: Cary Gross, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thanarajasingam G, Kluetz P, Bhatnagar V, Brown A, Cathcart-Rake E, Diamond M, Faust L, Fiero MH, Huntington S, Jeffery MM, Jones L, Noble B, Paludo J, Powers B, Ross JS, Ritchie JD, Ruddy K, Schellhorn S, Tarver M, Dueck AC, Gross C. Integrating 4 methods to evaluate physical function in patients with cancer (In4M): protocol for a prospective cohort study. BMJ Open. 2024 Jan 10;14(1):e074030. doi: 10.1136/bmjopen-2023-074030. PMID 38199641
- [Derived] Thanarajasingam G, Kluetz PG, Bhatnagar V, Brown A, Cathcart-Rake E, Diamond M, Faust L, Fiero MH, Huntington SF, Jeffery MM, Jones L, Noble BN, Paludo J, Powers B, Ross JS, Ritchie JD, Ruddy KJ, Schellhorn SE, Tarver ME, Dueck AC, Gross CP. Integrating 4 Measures to Evaluate Physical Function in Patients with Cancer (In4M): Protocol for a prospective study. medRxiv [Preprint]. 2023 Mar 9:2023.03.08.23286924. doi: 10.1101/2023.03.08.23286924. PMID 36945495

DOCUMENTS (1):
  • Informed Consent Form (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT05214144/ICF_000.pdf